CLINICAL TRIAL: NCT05037669
Title: Phase I Trial of Programmed Allogeneic CRISPR-edited T Cells (PACE) Gene Edited to Eliminate Endogenous TCR, HLA-class I and HLA-class II and Engineered to Express Anti-CD19 Chimeric Antigen Receptor (PACE CART19) in Patients With Relapsed Or Refractory CD19+ Leukemia and Lymphoma
Brief Title: Programmed Allogeneic CRISPR-edited T Cells Engineered to Express Anti-CD19 Chimeric Antigen Receptor (PACE CART19) in Patients With Relapsed Or Refractory CD19+ Leukemia and Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No available investigational product
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 27419
Record Dates: First submitted 2021-08-24; First posted 2021-09-08 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2022-03

CONDITIONS: Acute Lymphoblastic Leukemia; Chronic Lymphocytic Leukemia; Non Hodgkin Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Acute Lymphoblastic Leukemia (ALL) (Experimental): Adult patients aged >18 with relapsed or refractory B cell malignancies - Acute Lymphoblastic Leukemia (ALL)
  Interventions: Biological: PACE CART19
- Cohort B: Chronic Lymphocytic Leukemia (CLL) + Non-Hodgkin's Lymphoma (NHL) (Experimental): Adult patients aged >18 with relapsed or refractory B cell malignancies - Chronic Lymphocytic Leukemia (CLL) and Non-Hodgkin's Lymphoma (NHL).
  Interventions: Biological: PACE CART19

INTERVENTIONS:
Biological: PACE CART19 — PACE CART19 cells are allogeneic T cells transduced with a lentiviral vector to express an anti-CD19 scFv TCRz:41BB and electroporated to temporarily express the CRISPR/Cas9 RNA system resulting in beta-2 microglobulin (B2M), Class II Major Histocompatibility Complex Transactivator (CIITA) and TCR-α chain (TRAC) targeted disruption. PACE CART19 cells will be administered by IV infusion.

SUMMARY:
This is a Phase I trial to assess the safety and feasibility of administering pre-manufactured allogeneic T cells from healthy donors expressing CD19-targeting chimeric antigen receptors lacking expression of HLA class I, HLA class II molecules and endogenous TCR through CRISPR-mediated genome-editing of beta-2 microglobulin, CIITA and T cell receptor alpha chain, respectively. These cells are called PACE CART19 cells.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Documentation of CD19 expression on malignant cells

   a. ALL/CLL: At time of most recent relapse b. NHL: Within 6 months of physician-investigator confirmation of eligibility as long as there has been no intervening CD19 directed therapy since expression confirmed. Results outside of this window may be used, if there is no accessible tumor site and the subject did not receive intervening CD19 directed therapy since CD19 expression was confirmed.
3. Patients with relapsed disease after prior autologous or allogeneic SCT must meet the following criteria:

   a. Have no active GVHD and require no immunosuppression b. Are more than 6 months from transplant at the time of physician-investigator confirmation of eligibility
4. Adequate organ function defined as:

   1. Creatinine ≤ 1.6 mg/dl
   2. ALT/AST ≤ 3x upper limit of normal range
   3. Direct bilirubin ≤2.0 mg/dl, unless the subject has Gilbert's syndrome (≤3.0 mg/dl)
   4. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea, pulse oxygen > 92% on room air, and DLCO ≥ 40% (corrected for anemia)
   5. Left Ventricle Ejection Fraction (LVEF) ≥ 40% confirmed by ECHO/MUGA
5. Evidence of active disease. This could include circulating disease in the blood, disease in the bone marrow by standard morphology (or by MRD testing for ALL patients), or measurable disease per Lugano Criteria (NHL patients).
6. Male or female age ≥ 18 years.
7. ECOG Performance Status that is either 0 or 1.
8. Subjects of reproductive potential must agree to use acceptable birth control methods.
9. Disease-specific criteria:

   a. Cohort A i. Patients with relapsed or refractory B cell ALL which meets one of the following criteria:

<!-- -->

1. Relapsed or refractory B cell ALL with 2nd or greater relapse or refractory to 1st salvage as defined by:

   a. Recurrent disease in the blood or bone marrow identified morphologically, by immunohistochemistry or by Flow cytometry.

   b. Patients with extramedullary relapse only (no bone marrow involvement) will be eligible if disease response can be assessed radiographically, OR
2. Refractory B cell ALL as defined by:

   a. Failure to achieve remission (<5% bone marrow blasts) after 2 cycles of induction chemotherapy b. Patients that achieve morphologic remission but remain MRD+ after ≥2 cycles of induction chemotherapy, OR
3. Ph+ relapsed or refractory B cell ALL that is intolerant to or have failed a tyrosine kinase inhibitor therapy containing regimen.

ii. Patients with prior or current history of CNS3 disease* will be eligible only if CNS disease is responsive to therapy (at infusion, must meet criteria in Section 5.2) 1. *CNS disease definitions70:

a. CNS1 - no blasts seen on cytocentrifuge (CNS negative); b. CNS2 - total nucleated cell count <5x106/L, but blasts seen on cytocentrifuge; c. CNS3 - total nucleated cell count 5x106/L with blasts on cytocentrifuge and/or signs of CNS leukemia (i.e. cranial nerve palsy).

b. Cohort B (CLL) i. Patients must have relapsed/refractory disease after at least 2 prior lines of appropriate therapy, AND ii. Patients must have previously received, or be intolerant to an approved BTK inhibitor and venetoclax; unless a BTK inhibitor or venetoclax is contraindicated.

c. Cohort B (NHL)- With one of the following diagnoses: i. Diffuse Large B-cell Lymphoma

1. Patients with any of the following histologies:

   1. Diffuse large B-cell lymphoma (DLBCL), NOS

   i. Germinal center B-cell type ii. Activated B-cell type b. Primary cutaneous DLBCL, leg type c. Primary mediastinal (thymic) large B-cell lymphoma d. ALK+ large B-cell lymphoma e. High-grade B-cell lymphoma, with MYC and BCL2 and/or BCL6 rearrangements (i.e. "Double or Triple Hit") f. High-grade B-cell lymphoma, NOS
2. Patients must have relapsed after, or be ineligible for, prior CAR T cell therapy, and meet one of the following criteria:

   1. Relapsed/refractory disease after at least 2 prior lines of appropriate therapy and are ineligible for autologous stem cell transplant or commercial CAR T cell therapy.
   2. Relapse/refractory disease after autologous SCT.
   3. Relapsed/refractory disease after allogeneic SCT. ii. Large cell transformation of CLL (Richter's transformation)

1. Patients must be primary refractory or received at least 1 prior line of treatment.

iii. Follicular lymphoma 1. Patients who have received at least 2 prior lines of appropriate therapy (not including single agent monoclonal antibody therapy), AND 2. Progressed within 2 years after second or higher line of therapy. iv. Mantle cell lymphoma

1. Patients must have either failed or be ineligible for standard of care Tecartus™ (brexucabtagene autoleucel) or other investigational CAR T cell product; and
2. Patients must also meet one of the following criteria:

   1. Relapsed/refractory disease after at least 2 prior lines of appropriate therapy, including a BTK inhibitor. Single-agent monoclonal antibody therapy does not count towards prior lines of therapy.
   2. Relapsed/refractory disease after prior autologous SCT.
   3. Relapsed/refractory disease after prior allogeneic SCT..

Exclusion Criteria:

1. Active hepatitis B, active hepatitis C, or other active, uncontrolled infection.
2. Class III/IV cardiovascular disability according to the New York Heart Association Classification.
3. Clinically apparent arrhythmia or arrhythmias who are not stable on medical management within two weeks of physician-investigator confirmation of eligibility.
4. Active acute or chronic GVHD requiring systemic therapy.
5. Dependence on systemic steroids or immunosuppressant medications. For additional details regarding use of steroid and immunosuppressant medications.
6. Receipt of immune checkpoint inhibitors within 4 months prior to physician-investigator confirmation of eligibility.
7. CNS3 disease that is progressive on therapy, or with CNS parenchymal lesions.
8. Pregnant or nursing (lactating) women.
9. Patients with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system, and unrelated to their cancer or previous cancer treatment.
10. Active autoimmune disease requiring systemic immunosuppressive treatment equivalent to ≥ 10mg of prednisone. Patients with autoimmune neurologic diseases (such as MS) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2038-01 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events | 28 days
Time from consent to first PACE CART19 infusion. | 12 months
The number of subjects consented and treated and the number of subjects consented but never treated will be described. | 12 months

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 12 months
Best Overall Response (BOR) | 12 months
Overall Survival (OS) | 12 months
Event-free survival (EFS) | 12 Months
Duration of Response (DOR) | 12 Months
Kinetics of expansion, persistence and homing to marrow and other organs of infused cells by quantitative PCR. | 12 Months
Kinetics of expansion, persistence and homing to marrow and other organs of infused cells by flow cytometry. | 12 Months
Systemic soluble immune factors in serum before and after treatment, and during CRS. | 12 Months
Polychromatic flow cytometry-based assessment of leukemia and B cells, extent and duration of leukemic response | 12 Months
Use of Next-Generation Immunoglobulin heavy chain Sequencing (NGIS) to quantitate presence or absence of malignant B cells | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Frey, MD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided